CLINICAL TRIAL: NCT03571152
Title: Efficacy of the Use of Educational Videos for Caregivers of Patients in Subacute Phase of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Claudia Sanchez, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SIDISI: 101781
Record Dates: First submitted 2018-06-17; First posted 2018-06-27 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: Caregivers; Educational videos; Subacute phase
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Pre-experimental study design The level of practice and knowledge of the caregiver will be evaluated according to the video(s) corresponding to the session. Patient participation is expected for the evaluation of the caregiver's level of practice. After thirty minutes of use of the video, the level of practice and knowledge of the caregiver will be evaluated again for the same video. In each session this methodology will continue until the eighth video. At the end of all the videos, the level of satisfaction of the caregivers in relation to the videos will be evaluated.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational videos (Experimental): Subjects allocated in this arms will receive the educational videos.
  Interventions: Other: Educational videos

INTERVENTIONS:
Other: Educational videos — The level of practice and knowledge of the caregiver will be evaluated according to the video(s) corresponding to the session. Patient participation is expected for the evaluation of the caregiver's level of practice. After thirty minutes of use of the video, the level of practice and knowledge of the caregiver will be evaluated again for the same video. In each session this methodology will continue until the eighth video. At the end of all the videos, the level of satisfaction of the caregivers in relation to the videos will be evaluated.

SUMMARY:
Stroke is the second cause of death and third of disability in the adult population, By 2020 it is projected like the fourth cause of disability-adjusted life year (DALY) and by 2030 it is estimated that it will lead the global burden of morbidity from chronic noncommunicable diseases. As a consequence of stroke, patients show a certain degree of dependence and spend most of their time with a caregiver, especially since the subacute phase of the stroke. 80% of patients who survive have motor problems. The proper care during the first three months will significantly improve until 95% the patient rehabilitation. Caregivers have reported the need for information about clinical, prevention and treatment of stroke, like information about specific tasks of patient care, mobilizations, exercises, etc. Therefore, it is necessary to train and educate the caregivers in physical aspects of care, recovery and secondary prevention. However, oversaturated health systems, insufficient number of specialists, social inequity, limited coverage and speed of access to health services are factors that make difficult to educate caregivers. Studies have demonstrated that the Information Technology applied to health is a promising solution to educate and empower the patient, carer and family. For instance, the use of educational videos to improve the level of practice or knowledge of patients with chronic pain and chronic obstructive pulmonary disease. This project aims to evaluate the efficacy of the use of educational videos for caregivers of patients in subacute phase of stroke through of the change of the level of practice, knowledge and satisfaction.

DETAILED DESCRIPTION:
Sample size A sample size of 10 participants, it is possible to detect minimum differences of 10% to 20%, with standard deviations of 5% to 10%.

Statistical analysis plan The data collected will be entered into a database in Microsoft Excel, to be analyzed by the Epi Info statistical program. The qualitative variables will be analyzed by frequencies and percentages, the quantitative variables by arithmetic mean and standard deviation, some of them categorized for its interpretation. The bivariate analysis between two qualitative variables will be carried out using Fisher's exact test, the analysis between a qualitative variable and a quantitative one will be carried out through the Mann-Whitney U tests (non-normal distribution) and Student's t test (normal distribution). After the intervention, the level of practice and knowledge of the caregivers on the basic management of patients in the subacute phase of the stroke will generate a variable called "change of score", whose p-value should be less than 0.05.

Plan for missing data Due to the characteristics of the intervention, the investigators do not expect much loss to follow up patients after recruitment. However, all missing data will be reported as such.

ELIGIBILITY:
Inclusion Criteria:

* Familiar or known of patients in the subacute phase of ischemic stroke.
* Familiar or known of stable dependent patients with diagnosis of hemiplegia.
* Caregiver aged 18-65 years.

Exclusion Criteria:

* Caregiver with cognitive , severe auditory and/or visual problems.
* Caregiver of patients who do not collaborate due to their cognitive, neurological or psychiatric conditions.
* Caregiver of patients with comorbidities that affect mobility, such as other neurological disorders, orthopedic and/or traumatological alterations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Practice level | Before and after 30 minutes of watching each video the participant will be evaluated. This method will be used for the 8 videos developed. Therefore, there will be a change in the practice level.
  We will use the "evaluation form of the practice level", a check list with items that the caregiver should perform for the 8 activities represented in the 8 videos, for each activity a minimum of 4 items and a maximum of 9 items will be evaluated. The number of items for each activity is summed, so the total number of items is 49. Therefore, the minimum score is 0% (the caregiver performed 0% of items) and the maximum score is 100% (the caregiver performed 100% of items). The higher percentage represents a better result. This instrument will be review for experts, so the number of items could change.

SECONDARY OUTCOMES:
Knowledge level | Before and after 30 minutes of watching each video, the participant will be evaluated. This method will be used for the 8 videos developed. Therefore, there will be a change in the knowledge level.
  We will use the "evaluation form of the knowledge level", which was designed for the study, a questionnaire with one-answer questions related to 8 activities represented in the 8 videos, for each activity a minimum of 2 questions and a maximum of 4 questions will be evaluated. The number of questions for each activity is summed, so the total number of questions is 25. Therefore, the minimum score is 0% (the caregiver answered correctly 0% of questions) and the maximum score is 100% (the caregiver answered correctly 100% of questions). The higher percentage represents a better result. This instrument will be review for experts, so the number of questions could change.
Satisfaction level | After of watching all the videos, the participant will be evaluated. Minimum 1 video and maximum 3 videos will be evaluated per day. Therefore, minimum 3 days and maximum 8 days will be needed. The days will not be necessarily followed.
  We will use the "evaluation form of the satisfaction level", which was designed for the study, a questionnaire with 3 questions of Likert scale and 2 opened questions related to the 8 videos. Therefore, the results will be reported according to each question. This instrument will be review for experts, so this could change.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Sánchez Huamash, BSc, Principal Investigator
Locations (1):
- Universidad Cayetano Heredia, Lima, San Martín de Porres, Peru

IPD SHARING:
Plan to Share IPD: No
There is no plan description. No applicable.

REFERENCES:
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Vive-Larsen J, Stoier M, Olsen TS. Outcome and time course of recovery in stroke. Part I: Outcome. The Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 May;76(5):399-405. doi: 10.1016/s0003-9993(95)80567-2. PMID 7741608
- [Background] Kwakkel G, Kollen B, Lindeman E. Understanding the pattern of functional recovery after stroke: facts and theories. Restor Neurol Neurosci. 2004;22(3-5):281-99. PMID 15502272
- [Background] Karthikbabu S, Chakrapani M, Ganeshan S, Rakshith KC, Nafeez S, Prem V. A review on assessment and treatment of the trunk in stroke: A need or luxury. Neural Regen Res. 2012 Sep 5;7(25):1974-7. doi: 10.3969/j.issn.1673-5374.2012.25.008. PMID 25624827
- [Background] Duncan P, Studenski S, Richards L, Gollub S, Lai SM, Reker D, Perera S, Yates J, Koch V, Rigler S, Johnson D. Randomized clinical trial of therapeutic exercise in subacute stroke. Stroke. 2003 Sep;34(9):2173-80. doi: 10.1161/01.STR.0000083699.95351.F2. Epub 2003 Aug 14. PMID 12920254
- [Background] Di Monaco M, Trucco M, Di Monaco R, Tappero R, Cavanna A. The relationship between initial trunk control or postural balance and inpatient rehabilitation outcome after stroke: a prospective comparative study. Clin Rehabil. 2010 Jun;24(6):543-54. doi: 10.1177/0269215509353265. PMID 20511303
- [Background] Young ME, Lutz BJ, Creasy KR, Cox KJ, Martz C. A comprehensive assessment of family caregivers of stroke survivors during inpatient rehabilitation. Disabil Rehabil. 2014;36(22):1892-902. doi: 10.3109/09638288.2014.881565. Epub 2014 Jan 28. PMID 24467676
- See also: The role of caregiver involvement in upper-limb treatment in individuals with subacute stroke. — https://www.ncbi.nlm.nih.gov/pubmed/20592268